CLINICAL TRIAL: NCT06052319
Title: A Pilot Study to Assess the Engagement and Usefulness of Care4Today Digital Platform for Disease Management in Coronary Artery Disease/ Peripheral Artery Disease (CAD/PAD) Population
Brief Title: A Study to Assess the Engagement and Usefulness of Care4Today Digital Platform for Disease Management in Coronary Artery Disease (CAD) and/or Peripheral Artery Disease (PAD) Population
Acronym: IPACE-CVD
Status: Completed | Type: Observational
Sponsor: Janssen Scientific Affairs, LLC (Industry)
Collaborators: HCA Research Institute, LLC (Unknown)
Responsible Party: Sponsor
Other Study IDs: NOPRODPEA0001; NOPRODPEA0001 (Other: Janssen Scientific Affairs, LLC)
Record Dates: First submitted 2023-09-18; First posted 2023-09-25 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Coronary Artery Disease (CAD); Peripheral Artery Disease (PAD)
Keywords: Care4Today, Coronary Artery Disease, Peripheral Artery Disease, CAD, PAD
MeSH Terms: conditions — Coronary Artery Disease; Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with Coronary Artery Disease (CAD) or Peripheral Artery Disease (PAD) or Both: Participants with CAD or PAD or both will be directed to download the Care4Today® (C4T) Connect CAD-PAD mobile application on iPhone or Android device to assess engagement and usefulness of C4T in disease management for 3 months. No study drug and other treatment(s) will be provided as a part of this study. All aspects of treatment and clinical management of participants will continue to be in accordance with local clinical practice and applicable local regulations, and at the discretion of the participating physician.
  Interventions: Device: Care4Today® Connect CAD-PAD Mobile Application

INTERVENTIONS:
Device: Care4Today® Connect CAD-PAD Mobile Application — Participants will not receive any drug intervention in this study. Participants will use Care 4Today® Connect CAD-PAD mobile application for 3 months. The study will assess participant engagement and usefulness.

SUMMARY:
The purpose of this study is to assess the engagement and usefulness of Care4Today® Connect CAD-PAD digital platform in participants with coronary artery disease or peripheral artery disease (CAD or PAD).

ELIGIBILITY:
Inclusion Criteria:

* Must have a diagnosis of CAD and or PAD, who are on therapy or about to initiate therapy
* Own an iPhone or Android mobile device
* Have an active email account
* Must sign a participation agreement or informed consent form (ICF) allowing data collection in accordance with local requirements
* Willing to download and use Care4Today (C4T) CAD-PAD application (app)

Exclusion Criteria:

* Any cardiovascular conditions (for example, recent stroke, high bleeding risk, severe heart failure) or non-cardiovascular condition deemed as poor prognosis by the investigator and which may percent a patient from completing the study
* Unable to read or write the language used for the C4T (English, or Spanish if Spanish version is available)
* Visual or hearing impairment or mental disability that would preclude independent app use
* Patients currently using the C4T app prior to the signing of ICF

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include participants ages 40-90 diagnosed with coronary artery disease (CAD) or peripheral artery disease (PAD) or both.
Sampling Method: Non-Probability Sample
Enrollment: 277 (Actual)
Dates: Start 2023-11-29 (Actual); Primary Completion 2024-08-13 (Actual); Study Completion 2024-08-13 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Who use the Care4Today (C4T) Coronary Artery Disease-Peripheral Artery Disease (CAD-PAD) Application for at Least 10 Weeks During the 3-Month Study Period | Up to 3 months
  Percentage of participants (of those who onboarded the C4T CAD-PAD app) who use CAD-PAD the application for at least 10 weeks during the 3-month study period will be reported. The weekly app use is defined as using at least one component of the app once a week.
Percentage of Engaged Participants who Complete End of Study Survey with Satisfaction Response Score of Greater Than or Equal to (>=) 2 for at Least 3 Questions | Up to 3 months
  Percentage of engaged participants who complete end of study survey with satisfaction response score of >= 2 for at least 3 questions (out of 6 total questions) will be reported. Satisfaction survey consists of six questions in the end of study - each with 5 possible responses on a likert scale (1-5). The lowest possible response to any question is 1 =disagree and the highest possible response to any question is 5 = agree. Higher response on this scale represents more agreement or satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Scientific Affairs, LLC Clinical Trial, Study Director — Janssen Scientific Affairs, LLC
Locations (6):
- United States (6):
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - HCA Florida Memorial Hospital, Jacksonville, Florida
  - University of Florida Health Jacksonville, Jacksonville, Florida
  - The Kansas City Heart Rhythm Institute, Overland Park, Kansas
  - HCA Houston Healthcare Medical Center, Houston, Texas
  - Rio Grande Regional Hospital, McAllen, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lakkireddy D, Angiolillo DJ, Charlton-Ouw K, Jefferson B, Peeran S, Bisharat M, Ortega-Paz L, Harxhi A, Kaul S, Michaud E, Juan S, Woods B, Damaraju CV, Fontana G, Bonaca MP. Rationale and Design of a Study to Assess the Engagement and Usefulness of the Care4Today Connect Digital Health Application for Disease Management in Coronary Artery Disease and Peripheral Artery Disease (iPACE-CVD Study). Clin Cardiol. 2024 Dec;47(12):e70039. doi: 10.1002/clc.70039. PMID 39663755